CLINICAL TRIAL: NCT07237698
Title: A Study on the Effectiveness of Comprehensive Intervention Based on Specialized Physical Education Courses in the Prevention of Comorbidity Among Junior Middle School Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaoyan Wu (Other)
Responsible Party: Sponsor-Investigator, Xiaoyan Wu, Associate Researcher, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20250813
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Multimorbidity; Comorbidity; Common Diseases in Children and Adolescents; Myopia; Anxiety Symptoms; Depressive Symptoms; Overweight , Obesity
MeSH Terms: conditions — Myopia; Anxiety Disorders; Depression; Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group participated in regular physical education classes. (No Intervention)
- The intervention group participated in specialized physical education courses. (Experimental)
  Interventions: Other: The intervention group participated in specialized physical education courses.

INTERVENTIONS:
Other: The intervention group participated in specialized physical education courses. — Intervention Measures for This Study: During school hours, a portion of regular physical education classes will be replaced with specialized physical education courses jointly developed by the research team and school physical education teachers. These specialized courses aim to enhance the enjoyment of physical education, increase student participation, and consequently boost physical activity levels. The specialized physical education curriculum comprises five courses: darts, frisbee, flag football, handball, and orienteering. Students have one physical education class daily during their five-day school week. Routine physical education classes proceed as normal during school hours, ensuring both study groups complete one daily physical education class except under special circumstances. On weekdays, the intervention group replaces routine physical education classes with specialized physical education classes three days per week. These specialized classes are taught by dedicated physi
  Arms: The intervention group participated in specialized physical education courses.

SUMMARY:
Junior high school students are in a critical period of physical and mental development, currently facing two major health challenges: first, persistently high rates of myopia with a noticeable trend toward younger onset; second, the overlapping occurrence of common conditions such as overweight/obesity, spinal deformities, and psychological anxiety.Traditional physical education classes, characterized by limited content and insufficient targeting, struggle to address these issues. Multimorbidity of common diseases in children and adolescents refers to the coexistence of two or more common diseases or chronic health problems in the same individual.

Therefore, this study innovatively designed a specialized physical education curriculum integrating "exercise + health education," aiming to fill the gap in comprehensive prevention and control of common adolescent health conditions through traditional physical interventions.

This study systematically investigated the effects of a specialized physical education intervention program on myopia prevention and control, as well as the simultaneous prevention of multiple common health conditions (overweight/obesity, abnormal blood pressure, insufficient cardiorespiratory fitness, abnormal spinal curvature, anxiety symptoms, and depression symptoms) among junior high school students in China. The program was designed and implemented for students at a Chinese secondary school, ultimately aiming to provide a replicable school-based physical education intervention model for adolescent health promotion. The study strictly adhered to a randomized controlled design, employing multidimensional evaluation, long-term follow-up, and rigorous quality control to ensure scientific validity and reliability of the findings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who voluntarily participate in this study and whose parents or guardians voluntarily sign the informed consent form.
* Individuals capable of cooperating to complete measurements of all indicators throughout the entire intervention cycle.

Exclusion Criteria:

* Individuals with eye conditions such as glaucoma, strabismus, or anisometropia.
* Wearers of orthokeratology lenses.
* Individuals who have undergone refractive surgery.
* Individuals who have taken weight-loss medications or undergone weight-loss surgery.
* Individuals with obesity caused by endocrine disorders or medication side effects.
* Individuals with mental health disorders.
* Individuals currently taking medications for mental health disorders.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Multimorbidity of common diseases | baseline、"through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: Undecided